CLINICAL TRIAL: NCT02850146
Title: 18F-AV-1451 PET Imaging in Participants Enrolled in the LEARN Study
Acronym: LEARN-Tau
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Alzheimer's Therapeutic Research Institute (Other); Alzheimer's Association (Other); Avid Radiopharmaceuticals (Industry)
Responsible Party: Principal Investigator, Paul Aisen, Director, Alzheimer's Therapeutic Research Institute, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A17; 15-338729 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cognition Disorders
Keywords: tau; cognition; longitudinal; cognitive decline; observational; imaging
MeSH Terms: conditions — Cognition Disorders; Pick Disease of the Brain; Cognitive Dysfunction | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-AV-1451 (Experimental): 50 individuals who are cognitively normal, older, Aβ not elevated and enrolled in the LEARN study will undergo 18F-AV-1451 imaging procedures at 4 time points over a 4.5 year period.
  Interventions: Drug: 18F-AV-1451

INTERVENTIONS:
Drug: 18F-AV-1451

SUMMARY:
Approximately 50 participants enrolled in the LEARN study (NCT02488720) will be enrolled in the LEARN-Tau study. The study designed to evaluate the imaging characteristics of 18F-AV-1451 in participants enrolled in the LEARN study and to expand the safety database of 18F-AV-1451.

The study will run in parallel to the LEARN study. In this study, participants will undergo up to four (4) 18F-AV-1451 PET scans over a 4.5 year period. Imaging visits will occur at the throughout the participant's participation in the LEARN study (corresponding to LEARN Visit 1, between Visit 4 and 6, Visit 8, and Visit 11).

The LEARN-Tau study will (1) look at change in the amount of tau protein in the brain over time, measured by the 18F-AV-1451 PET scan, (2) see if tau protein in the brain of older individuals is associated with memory problems and (3) evaluate the safety of 18F-AV-1451 and any side effects that might be associated with it.

Site investigators, participants, and study partners will not be informed of the results of the 18F-AV-1451 PET scan results as they relate to the study; however, any findings that may be of potential medical concern will be provided for appropriate follow-up.

ELIGIBILITY:
Participants should meet inclusion and exclusion criteria for the LEARN study, and in addition:

Inclusion Criteria:

* Male or female that have consented and are currently enrolled in the LEARN protocol;
* Participants who sign an IRB approved informed consent form prior to any study procedure; and
* Participants who in the opinion of the investigator can tolerate the PET scan procedures.

Exclusion Criteria:

* Has any condition that, in the investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with analysis of the data. (For example, participants with chronic back pain might not be able to lie still during the scanning procedures.);
* Has abnormal findings on physical examination or laboratory screening tests that suggest the participant might have a condition that could, in the opinion of the investigator, affect his or her response to the radiopharmaceutical and related testing procedures;
* Is deemed likely to be unable to perform all of the imaging procedures for any reason;
* Has a history of risk factors for torsades de pointes, including clinically significant findings on ECG, or is taking medications known to prolong QT interval such as citalopram ≥ 40 mg/day, disopyramide, dofetilide, ibutilide, procainamide, quinidine, sotalol, or bepridil; A list of restricted medications will be provided.
* Are females of childbearing potential (extremely unlikely in the LEARN eligible population ages 65 to 85) who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception. Females of childbearing potential must not be pregnant (negative serum or urine β-hCG at the time of screening and negative serum or urine β-hCG on imaging day) or breastfeeding at screening. Females must agree to avoid becoming pregnant, and both females and males must agree to refrain from sexual activity or to use reliable contraceptive methods for 24 hours following administration of 18F-AV-1451 Injection; Males with female partners who are pregnant or of childbearing potential must agree to refrain from sexual activity for 24 hours following administration of 18F-AV-1451 Injection. Additionally, males must agree not to donate sperm for 24 hours following administration of 18F-AV-1451 Injection;
* Has hypersensitivity to 18F-AV-1451 or any of its excipients.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-08; Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Rate of change of tau deposition as measured by 18F-AV-1451 | 3 years
Change in tau deposition as measured by 18F-AV-1451 standardized uptake value ratio (SUVR) from the baseline scan | Baseline, 84 weeks, 168 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reisa Sperling, MD, Study Director — Center for Alzheimer Research and Treatment Brigham and Women's Hospital
Locations (7):
- United States (7):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - Bioclinica Research North, The Villages, Florida
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Butler Hospital Memory and Aging Program, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chien DT, Bahri S, Szardenings AK, Walsh JC, Mu F, Su MY, Shankle WR, Elizarov A, Kolb HC. Early clinical PET imaging results with the novel PHF-tau radioligand [F-18]-T807. J Alzheimers Dis. 2013;34(2):457-68. doi: 10.3233/JAD-122059. PMID 23234879
- [Background] Duyckaerts C, Brion JP, Hauw JJ, Flament-Durand J. Quantitative assessment of the density of neurofibrillary tangles and senile plaques in senile dementia of the Alzheimer type. Comparison of immunocytochemistry with a specific antibody and Bodian's protargol method. Acta Neuropathol. 1987;73(2):167-70. doi: 10.1007/BF00693783. PMID 2440224
- [Background] Nelson PT, Alafuzoff I, Bigio EH, Bouras C, Braak H, Cairns NJ, Castellani RJ, Crain BJ, Davies P, Del Tredici K, Duyckaerts C, Frosch MP, Haroutunian V, Hof PR, Hulette CM, Hyman BT, Iwatsubo T, Jellinger KA, Jicha GA, Kovari E, Kukull WA, Leverenz JB, Love S, Mackenzie IR, Mann DM, Masliah E, McKee AC, Montine TJ, Morris JC, Schneider JA, Sonnen JA, Thal DR, Trojanowski JQ, Troncoso JC, Wisniewski T, Woltjer RL, Beach TG. Correlation of Alzheimer disease neuropathologic changes with cognitive status: a review of the literature. J Neuropathol Exp Neurol. 2012 May;71(5):362-81. doi: 10.1097/NEN.0b013e31825018f7. PMID 22487856
- [Background] Xia CF, Arteaga J, Chen G, Gangadharmath U, Gomez LF, Kasi D, Lam C, Liang Q, Liu C, Mocharla VP, Mu F, Sinha A, Su H, Szardenings AK, Walsh JC, Wang E, Yu C, Zhang W, Zhao T, Kolb HC. [(18)F]T807, a novel tau positron emission tomography imaging agent for Alzheimer's disease. Alzheimers Dement. 2013 Nov;9(6):666-76. doi: 10.1016/j.jalz.2012.11.008. Epub 2013 Feb 12. PMID 23411393
- See also: Alzheimer's Therapeutic Research Institute — https://keck.usc.edu/atri/research/studies/
- See also: Alzheimer's Association — http://www.alz.org/
- See also: Avid Radiopharmaceuticals — http://www.avidrp.com/